CLINICAL TRIAL: NCT02693743
Title: Repetitive Transcranial Magnetic Stimulation as Treatment for Acute Suicidality in Adult Patients
Acronym: rTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated early due to slow accrual or other non-safety related issues
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 203818
Record Dates: First submitted 2016-02-12; First posted 2016-02-29 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2020-04

CONDITIONS: Suicidal Ideation
Keywords: suicidality; rTMS; suicide ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active rTMS (Active Comparator): Repetitive Transcranial Magnetic Stimulation (rTMS) will be delivered to the left PFC, deﬁned as a location 6 cm (cm) anterior to the right hand motor thumb area. A research nurse will deliver the treatments. rTMS will be delivered with a ﬁgure-eight coil at 120% motor threshold, 10 Hertz (Hz), 5 s (s) train duration, 20 s intertrain interval for 50 min (6000 pulses) 3 times daily for 3 days (total 9 sessions, 54,000 stimuli).
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham rTMS (Sham Comparator): Parameters for sham Repetitive Transcranial Magnetic Stimulation (rTMS) are identical to those for active stimulation except that aluminum plate blocks the propagation of a magnetic field. The sound and physical sensation is the same as with the active coil while been biologically inactive.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — A Neurostar TMS Therapy System and Neurostar XPLOR coil system (Neuronetics, Malvern, Pennsylvania) will be used to deliver stimulation.

SUMMARY:
Suicide was responsible for almost 40,000 deaths in 2011 in America. It is still singularly difficult to predict who is going to commit suicide and how to establish adequate interventions. Growing evidence supports the view that suicide is associated with poor decision making. Suicide is hypothesized to be triggered by stressful situations that create overwhelming psychological pain in an individual who chooses to terminate his/her own life, disregarding all future consequences. We have previously demonstrated rewarding impulsive choice common to both recent suicide attempters and suicidal depressed patients (1). Consistent with these findings, we hypothesize that high frequency repetitive transcranial magnetic stimulation (rTMS) of the left prefrontal cortex will improve impulsive response tendencies as measured by the delay discounting procedure, and this in turn will be associated with a faster resolution of suicidal ideation. To these effects we will be using a randomized control trial of rTMS in adult inpatients at the Psychiatric Research Institute (PRI) hospitalized for acute suicidality. At the conclusion of these studies, we will have tested the value of decision making in the development of suicide ideation and behavior, as well as piloted the use of rTMS in the treatment of these patients.

DETAILED DESCRIPTION:
The proposed study seeks to improve the prevention of suicide by advancing our understanding of the neurobiology of suicide by using a randomized control trial of repetitive transcranial magnetic stimulation (rTMS) as a hypothesis driven intervention for acute suicidality. In 2010 suicide was responsible for more than 38,364 deaths in the United States and 447 in the state of Arkansas (CDC, 2012). Suicide represents the 10th leading cause of death in this country, and claims more deaths than chronic liver disease, hypertension, Parkinson's disease or homicide. Furthermore, suicide consequences extend beyond the termination of an individual's life to impact those that are left behind. These statistics are far more alarming because they are believed to be underestimates, with substantial numbers of suicides and suicide attempts undetected or misclassified. The high and rising prevalence of suicide is complicated by the clinical challenge of identifying those patients at highest risk for suicide. A variety of biological, psychological and social risk factors for suicide have been identified. However, we currently lack reliable predictors of suicide risk and must rely heavily upon self-report and clinical judgment. Thus, it remains singularly difficult to predict who is going to commit suicide. Therefore, there is an urgent unmet need to develop effective early detection methods and treatments for high-risk populations.

Suicide has been described as "a permanent solution to a temporary problem" (Buchwald, 2006), reflecting the view that suicide is the result of poor decision making. The strongest biological finding in suicide research is the association with reduced serotonergic neurotransmission, particularly within the ventromedial prefrontal cortex (VMPFC) (Mann, 2003). This deficit in serotonergic neurotransmission is thought to impair cognition, predisposing patients to become more impulsive, rigid in their thinking, and poorer decision makers. Decisions during depressed states are tainted by negative affect and distorted negative cognitions (Martin-Soelch, 2009). However, suicide has been associated with cognitive impairments that go beyond those of depression. Asymptomatic patients with a history of suicide attempts exhibit significant cognitive deficits suggestive of generalized prefrontal cortex (PFC) dysfunction (Raust et al, 2007; Westheide et al, 2008), and corollary disruptions in risk assessment (Martino et al, 2010). Poor inhibition is found in suicide attempters when compared with patients with only suicidal ideation (Burton et al, 2011), and greater cognitive impairments are found in depressed patients with suicidal ideation compared to those without it (Dombrovski et al, 2010). It is possible that cognitive deficits may be specific to suicidal behavior rather than to any comorbid or specific psychiatric diagnosis because this observation holds true for suicidal patients with depression, bipolar disorder, and even temporal lobe epilepsy. However, most of these studies were performed in symptom-free patients, often months or years after the presence of suicidal ideation or behavior. In a previous report (Cáceda et al, 2014) we demonstrated that inability to delay gratification (choosing smaller immediate rewards over larger delayed rewards) is shared by both recent suicide attempters and depressed patients with suicidal ideation. On a follow up assessment, 5-10 days after the suicide attempt, reduction of suicidal ideation and intent was correlated with decreased symptoms of depression and recovery of delayed gratification impairments (Cáceda et al, 2014). These data are congruent with the hypothesis that stressful situations in combination with a biological and psychological predisposition may create a critical climate of overwhelming psychological pain in an individual who chooses an impulsive escapist strategy to terminate his/her own life discounting all future outcomes (Vohs et al, 2002). However, the underlying neural mechanisms remain unknown and therefore not amenable to therapeutic interventions.

TMS is a noninvasive method to cause depolarization or hyperpolarization in the neurons in the brain using electromagnetic induction to induce weak electric currents using a rapidly changing magnetic field. TMS is a novel intervention developed in the field of neurology that has been used in the treatment of patients suffering from migraine, stroke, Parkinson's disease, tinnitus and depression. In healthy subjects, high frequency rTMS over the left DLPFC has been shown to alter impulsive choice behavior (to decrease delay discounting) in healthy individuals and in smokers (Sheffer et al, 2013). On the other hand, a trial of TMS by one of the leaders in the field has shown it to be safe and well tolerated in recent suicide attempters suffering from depression with comorbid post-traumatic stress disorder and traumatic brain injury (George et al, 2014).

Dr. Mennemeier, the director of the Transcranial Magnetic Stimulation Laboratory in the Center for Translational Neuroscience has been using repetitive transcranial magnetic stimulation (rTMS) to understand and treat phantom sound perception in subjects with tinnitus and to examine risky choices and impulsive behaviors using delay discounting in smokers. We propose to replicate a randomized controlled trial of rTMS over 3 days in a sample of well characterized acutely suicidal inpatients.

Our overall hypothesis is that 10 Hertz rTMS of the left dorsolateral prefrontal cortex (DLPFC) will correct impulsive choice behavior deficits found in acutely suicidal patients that in turn will translate into faster resolution of acute suicidal ideation. The current proposal will expand our understanding of the neurobiology of suicidal behavior by examining a potential neurocognitive mechanism of acute suicidality and test the value of rTMS as intervention for acute suicidal behavior. The current proposal will utilize behavioral assessments and rTMS in a randomized controlled trial in a group of adult patients hospitalized: a) following a recent suicide attempt with persistent suicidal ideation, or b) for severe suicidal ideation (n=20). Specifically, we propose:

Specific Aim 1. Determine the safety of repetitive transcranial magnetic stimulation (rTMS) in depressed patients with severe suicidal ideation.

Hypothesis 1: Given studies of rTMS for clinical depression, the investigators predict that rTMS in patients with severe suicidal ideation will be well tolerated and not associated with significant side effects.

Specific Aim 2. Determine the effect of rTMS on delay discounting on depressed patients with severe suicidal ideation.

Hypothesis 2: In depressed patients with severe suicidal ideation the rTMS active will reduce impulsive choice behavior (measured as delay discounting) compared with the non-treatment group.

Specific Aim 3. Determine the effect of rTMS on suicidal ideation on depressed patients with severe suicidal ideation.

Hypothesis 3.1: In depressed patients who had recently attempt suicide the rTMS active group will reduce suicidal ideation severity (measured by the Beck Scale for Suicidal Ideation) compared with the non-treatment group.

Hypothesis 3.2: Suicidal ideation in depressed patients who recently attempt suicide will vary in function of delay discounting.

Specific Aim 4. Identification of biomarkers of positive response to rTMS in depressed patients with severe suicidal ideation.

Hypothesis 4: A composite of serum hormonal and inflammatory markers will predict positive response to rTMS in depressed patients with severe suicidal ideation

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years, of all races and ethnicities;
* Admitted voluntarily to the adult psychiatric inpatient at PRI;
* Suffering from a current depressive episode
* Reason for hospitalization should be a recent suicide attempt or suicidal ideation
* Current severe suicidal ideation defined by a score >7 on the Beck Scale for Suicidal Ideation
* Ability to read, write and speak English.

Exclusion Criteria:

* History of dementia, neurovascular or neurodegenerative conditions
* Physical disabilities that prohibit task performance (such as blindness or deafness)
* Choosing to opt out of the research study.
* Additional exclusion criteria for TMS include the following:

  * a personal history or 1st degree relative with history of epilepsy;
  * a personal history of head injury, aneurysm, stroke, previous cranial neurosurgery, neurological, or migraines;
  * recent use of cocaine or alcohol;
  * ferromagnetic metal implants in the head or neck, active or inactive implants(including device leads), deep brain stimulators, cochlear implants or vagus nerve stimulators;
  * a pacemaker;
  * pregnancy (or the possibility of pregnancy);
  * Medications that lower seizure threshold (bupropion or tricyclic antidepressants, such as thorazine, clozapine, amitriptyline, amoxapine, Norpramin, Sinequan, Tofranil, Pamelor, Vivactil, or Surmontil). Other antidepressant and antipsychotic medications have been deemed exhibit a relatively low seizurogenic potential (Pisani et al. 2002).
  * Patients taking a medication for weight loss and depression called bupropion (Wellbutrin) they will be excluded because it may increase the likelihood of experiencing a seizure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro L Delgado, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caceda R, Durand D, Cortes E, Prendes-Alvarez S, Moskovciak T, Harvey PD, Nemeroff CB. Impulsive choice and psychological pain in acutely suicidal depressed patients. Psychosom Med. 2014 Jul-Aug;76(6):445-51. doi: 10.1097/PSY.0000000000000075. PMID 24988311
- [Background] Heins SE, Crifasi CK. Distinctive injury deaths: the role of environment, policy and measurement across states. Inj Prev. 2016 Aug;22(4):247-52. doi: 10.1136/injuryprev-2015-041833. Epub 2016 Jan 24. PMID 26804777
- [Background] Buchwald A. Too soon to say goodbye. 1st ed. New York: Random house; 2006.
- [Background] Mann JJ. Neurobiology of suicidal behaviour. Nat Rev Neurosci. 2003 Oct;4(10):819-28. doi: 10.1038/nrn1220. No abstract available. PMID 14523381
- [Background] Martin-Soelch C. Is depression associated with dysfunction of the central reward system? Biochem Soc Trans. 2009 Feb;37(Pt 1):313-7. doi: 10.1042/BST0370313. PMID 19143654
- [Background] Westheide J, Quednow BB, Kuhn KU, Hoppe C, Cooper-Mahkorn D, Hawellek B, Eichler P, Maier W, Wagner M. Executive performance of depressed suicide attempters: the role of suicidal ideation. Eur Arch Psychiatry Clin Neurosci. 2008 Oct;258(7):414-21. doi: 10.1007/s00406-008-0811-1. Epub 2008 Mar 11. PMID 18330667
- [Background] Raust A, Slama F, Mathieu F, Roy I, Chenu A, Koncke D, Fouques D, Jollant F, Jouvent E, Courtet P, Leboyer M, Bellivier F. Prefrontal cortex dysfunction in patients with suicidal behavior. Psychol Med. 2007 Mar;37(3):411-9. doi: 10.1017/S0033291706009111. Epub 2006 Oct 19. PMID 17049103
- [Background] Martino DJ, Strejilevich SA, Torralva T, Manes F. Decision making in euthymic bipolar I and bipolar II disorders. Psychol Med. 2011 Jun;41(6):1319-27. doi: 10.1017/S0033291710001832. Epub 2010 Sep 22. PMID 20860871
- [Background] Burton CZ, Vella L, Weller JA, Twamley EW. Differential effects of executive functioning on suicide attempts. J Neuropsychiatry Clin Neurosci. 2011 Spring;23(2):173-9. doi: 10.1176/jnp.23.2.jnp173. PMID 21677246
- [Background] Dombrovski AY, Clark L, Siegle GJ, Butters MA, Ichikawa N, Sahakian BJ, Szanto K. Reward/Punishment reversal learning in older suicide attempters. Am J Psychiatry. 2010 Jun;167(6):699-707. doi: 10.1176/appi.ajp.2009.09030407. Epub 2010 Mar 15. PMID 20231320
- [Background] Vohs KD, Baumeister R. Escaping the self consumes regulatory resources: a self-regulatory model of suicide. Suicide Science. 2002:33-41.
- [Background] Sheffer CE, Mennemeier M, Landes RD, Bickel WK, Brackman S, Dornhoffer J, Kimbrell T, Brown G. Neuromodulation of delay discounting, the reflection effect, and cigarette consumption. J Subst Abuse Treat. 2013 Aug;45(2):206-14. doi: 10.1016/j.jsat.2013.01.012. Epub 2013 Mar 18. PMID 23518286
- [Background] George MS, Raman R, Benedek DM, Pelic CG, Grammer GG, Stokes KT, Schmidt M, Spiegel C, Dealmeida N, Beaver KL, Borckardt JJ, Sun X, Jain S, Stein MB. A two-site pilot randomized 3 day trial of high dose left prefrontal repetitive transcranial magnetic stimulation (rTMS) for suicidal inpatients. Brain Stimul. 2014 May-Jun;7(3):421-31. doi: 10.1016/j.brs.2014.03.006. Epub 2014 Mar 19. PMID 24731434
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Hamilton M. Diagnosis and rating of anxiety. The British journal of psychiatry : the journal of mental science. 1969;3:76-9.
- [Background] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082
- [Background] Beck AT. Beck Hopelessness Scale. The Psychological Corporation; 1988.
- [Background] Kirby KN, Petry NM, Bickel WK. Heroin addicts have higher discount rates for delayed rewards than non-drug-using controls. J Exp Psychol Gen. 1999 Mar;128(1):78-87. doi: 10.1037//0096-3445.128.1.78. PMID 10100392
- [Background] Owen AM, McMillan KM, Laird AR, Bullmore E. N-back working memory paradigm: a meta-analysis of normative functional neuroimaging studies. Hum Brain Mapp. 2005 May;25(1):46-59. doi: 10.1002/hbm.20131. PMID 15846822
- [Background] Keilp JG, Gorlyn M, Russell M, Oquendo MA, Burke AK, Harkavy-Friedman J, Mann JJ. Neuropsychological function and suicidal behavior: attention control, memory and executive dysfunction in suicide attempt. Psychol Med. 2013 Mar;43(3):539-51. doi: 10.1017/S0033291712001419. Epub 2012 Jul 10. PMID 22781400
- [Background] REITAN RM. The relation of the trail making test to organic brain damage. J Consult Psychol. 1955 Oct;19(5):393-4. doi: 10.1037/h0044509. No abstract available. PMID 13263471
- [Background] Pridmore S, Fernandes Filho JA, Nahas Z, Liberatos C, George MS. Motor threshold in transcranial magnetic stimulation: a comparison of a neurophysiological method and a visualization of movement method. J ECT. 1998 Mar;14(1):25-7. PMID 9661090
- [Background] Mishory A, Molnar C, Koola J, Li X, Kozel FA, Myrick H, Stroud Z, Nahas Z, George MS. The maximum-likelihood strategy for determining transcranial magnetic stimulation motor threshold, using parameter estimation by sequential testing is faster than conventional methods with similar precision. J ECT. 2004 Sep;20(3):160-5. doi: 10.1097/00124509-200409000-00007. PMID 15343000
- [Background] Borckardt JJ, Nahas Z, Koola J, George MS. Estimating resting motor thresholds in transcranial magnetic stimulation research and practice: a computer simulation evaluation of best methods. J ECT. 2006 Sep;22(3):169-75. doi: 10.1097/01.yct.0000235923.52741.72. PMID 16957531
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossi S, De Capua A, Ulivelli M, Bartalini S, Falzarano V, Filippone G, Passero S. Effects of repetitive transcranial magnetic stimulation on chronic tinnitus: a randomised, crossover, double blind, placebo controlled study. J Neurol Neurosurg Psychiatry. 2007 Aug;78(8):857-63. doi: 10.1136/jnnp.2006.105007. Epub 2007 Feb 21. PMID 17314192
- [Background] Langguth B, de Ridder D, Dornhoffer JL, Eichhammer P, Folmer RL, Frank E, Fregni F, Gerloff C, Khedr E, Kleinjung T, Landgrebe M, Lee S, Lefaucheur JP, Londero A, Marcondes R, Moller AR, Pascual-Leone A, Plewnia C, Rossi S, Sanchez T, Sand P, Schlee W, Pysch D, Steffens T, van de Heyning P, Hajak G. Controversy: Does repetitive transcranial magnetic stimulation/ transcranial direct current stimulation show efficacy in treating tinnitus patients? Brain Stimul. 2008 Jul;1(3):192-205. doi: 10.1016/j.brs.2008.06.003. Epub 2008 Jul 1. PMID 20633385
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Pascual-Leone A, Houser CM, Reese K, Shotland LI, Grafman J, Sato S, Valls-Sole J, Brasil-Neto JP, Wassermann EM, Cohen LG, et al. Safety of rapid-rate transcranial magnetic stimulation in normal volunteers. Electroencephalogr Clin Neurophysiol. 1993 Apr;89(2):120-30. doi: 10.1016/0168-5597(93)90094-6. PMID 7683602
- [Background] Grafman J, Pascual-Leone A, Alway D, Nichelli P, Gomez-Tortosa E, Hallett M. Induction of a recall deficit by rapid-rate transcranial magnetic stimulation. Neuroreport. 1994 May 9;5(9):1157-60. doi: 10.1097/00001756-199405000-00034. PMID 8080978
- [Background] Flitman SS, Grafman J, Wassermann EM, Cooper V, O'Grady J, Pascual-Leone A, Hallett M. Linguistic processing during repetitive transcranial magnetic stimulation. Neurology. 1998 Jan;50(1):175-81. doi: 10.1212/wnl.50.1.175. PMID 9443476
- [Background] Pascual-Leone A, Gates JR, Dhuna A. Induction of speech arrest and counting errors with rapid-rate transcranial magnetic stimulation. Neurology. 1991 May;41(5):697-702. doi: 10.1212/wnl.41.5.697. PMID 2027485
- [Background] Counter SA, Borg E, Lofqvist L, Brismar T. Hearing loss from the acoustic artifact of the coil used in extracranial magnetic stimulation. Neurology. 1990 Aug;40(8):1159-62. doi: 10.1212/wnl.40.8.1159. PMID 2381522
- [Background] Mennemeier M, Chelette KC, Allen S, Bartel TB, Triggs W, Kimbrell T, Crew J, Munn T, Brown GJ, Dornhoffer J. Variable changes in PET activity before and after rTMS treatment for tinnitus. Laryngoscope. 2011 Apr;121(4):815-22. doi: 10.1002/lary.21425. Epub 2011 Feb 1. PMID 21287564
- [Background] Mennemeier M, Chelette KC, Myhill J, Taylor-Cooke P, Bartel T, Triggs W, Kimbrell T, Dornhoffer J. Maintenance repetitive transcranial magnetic stimulation can inhibit the return of tinnitus. Laryngoscope. 2008 Jul;118(7):1228-32. doi: 10.1097/MLG.0b013e318170f8ac. PMID 18475211
- [Background] Mennemeier M, Triggs W, Chelette K, Woods A, Kimbrell T, Dornhoffer J. Sham Transcranial Magnetic Stimulation Using Electrical Stimulation of the Scalp. Brain Stimul. 2009 Jul 1;2(3):168-173. doi: 10.1016/j.brs.2009.02.002. PMID 20160893
- [Background] Smith JA, Mennemeier M, Bartel T, Chelette KC, Kimbrell T, Triggs W, Dornhoffer JL. Repetitive transcranial magnetic stimulation for tinnitus: a pilot study. Laryngoscope. 2007 Mar;117(3):529-34. doi: 10.1097/MLG.0b013e31802f4154. PMID 17334317
- [Background] Roth BJ, Pascual-Leone A, Cohen LG, Hallett M. The heating of metal electrodes during rapid-rate magnetic stimulation: a possible safety hazard. Electroencephalogr Clin Neurophysiol. 1992 Apr;85(2):116-23. doi: 10.1016/0168-5597(92)90077-o. PMID 1373364
- [Background] Pascual-Leone A. Handbook of transcranial magnetic stimulation. London New York, NY: Arnold ; Oxford University Press distributor; 2002.
- [Background] Niehaus L, Hoffmann KT, Grosse P, Roricht S, Meyer BU. MRI study of human brain exposed to high-dose repetitive magnetic stimulation of visual cortex. Neurology. 2000 Jan 11;54(1):256-8. doi: 10.1212/wnl.54.1.256. PMID 10636165

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subject did not receive TMS due to technical difficulties with the equipment. Subject was withdrawn from the study by PI
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Beck Scale for Suicidal Ideation
Description: Change in suicidal ideation between baseline assessment and following 3 day TMS trial.
Time Frame: Within the 3 days of the TMS trial.
Population: No outcome measures were taken, subject did not receive TMS, due to technical difficulties. Subject was withdrawn by PI
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: There is no time frame for adverse events because none were reported. Subject was withdrawn from study and did not receive TMS.
Description: There is no adverse event information. Subject did not complete study.
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02693743/Prot_SAP_004.pdf